CLINICAL TRIAL: NCT05938803
Title: Community-Based Accompaniment for Adolescents Transitioning to Adult HIV Care in Urban Peru: an Evaluation of the "PASEO" Intervention
Brief Title: PASEO Intervention for Adolescents Transitioning to Adult HIV Care in Urban Peru
Acronym: PASEO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University Faculty of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Molly Franke, Professor of Global Health and Social Medicine, Harvard University Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01MH131414 (NIH); R01MH131414 (NIH)
Record Dates: First submitted 2023-06-13; First posted 2023-07-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: Adolescence; Community-based accompaniment; Retention; Antiretroviral treatment; Social support; Mental health; Treatment support; Adherence
MeSH Terms: conditions — HIV Infections; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (No Intervention): Participants randomized to the control arm of the study will receive a modestly enhanced standard of care. Specifically, they will receive HIV transition information in the form of a paper brochure and/or a video link, and a package of supplies (i.e., a pillbox, a folder to store medical documents). Participants will undergo depression and substance use screening and will be referred as needed.
- Intervention arm (Experimental): Participants randomized to the intervention arm of the study will receive a modestly enhanced standard of care. Specifically, they will receive HIV transition information in the form of a paper brochure and/or a video link, and a package of supplies (i.e., a pillbox, a folder to store medical documents). Participants will undergo depression and substance use screening and will be referred as needed. Participants allocated to this group will also receive the PASEO intervention.
  Interventions: Behavioral: PASEO

INTERVENTIONS:
Behavioral: PASEO — The intervention consists of community-based accompaniment intervention aimed at facilitating the transition to adult HIV care for adolescents living with HIV in Lima, Peru.The intervention includes the following activities: health systems navigation and accompaniment to clinic visits, monthly check-ins with an entry-level health worker, social support provided through peer support groups, education sessions, resolution of acute needs, and individualized adherence support.
  Arms: Intervention arm

SUMMARY:
This study is an evaluation of an intervention (nicknamed "PASEO") that aims to facilitate the transition to adult HIV care for adolescents living with HIV in Lima, Peru. The intervention consists of health systems navigation and accompaniment, monthly check-ins with a lay health worker, enhanced social support provided through peer support groups, education sessions, mental health screening and referral, resolution of acute needs, and individualized adherence support.

The study is a two-arm 1:1 randomized evaluation to determine the short- and long-term (i.e., post-intervention) efficacy of the PASEO intervention with regard to retention with viral load suppression as well as other indicators of well-being. The cumulative incidence of unsuccessful transition at 12- and 24-months will be compared. The cost and cost-effectiveness of the study intervention in terms of cost per additional successful transition achieved will be estimated. Data on implementation considerations essential for uptake, sustainability, and successful adoption by the public sector will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent or young person living with HIV and aware of diagnosis
* 14 to 21 years of age (may be increased to 23 to meet recruitment targets)
* Currently taking or eligible for ART at a participating facility
* Scheduled to transition to adult care or previous unsuccessful transition to adult care
* Willing to participate regardless of the study arm to which they will be assigned
* Able and willing to provide written informed consent

Exclusion Criteria:

* Living outside of Lima province
* Participation in the PASEO pilot study
* Current enrollment in another research study
* Having any condition (social or medical) which the study team considers would make participation unsafe

Ages: 14 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Unsuccessful transition | 12 months
  Number of people who experience death, loss to follow-up or unsuppressed viral load >200 copies/mL
Unsuccessful transition | 24 months
  Number of people who experience death, loss to follow-up or unsuppressed viral load >200 copies/mL

SECONDARY OUTCOMES:
HIV-related death or loss to follow-up | within 12 and 24 months
  Time to HIV-related death or loss to follow-up
Clinic visit attendance | 12 and 24 months
  Number of scheduled visits attended, among those retained
CD4 cell count | 12 and 24 months
  Change in CD4 cell count from baseline
Self-efficacy | 6, 9, 12, 24 months
  Change in self-efficacy (assessed using the NIH toolbox) from baseline
Transition readiness | 6, 9, 12, 24 months
  Change in transition readiness (assessed using the Am I on TRAC and Got Transitions questionnaires) from baseline
Perceived social support | 6, 9, 12, 24 months
  Change in social support (assessed using the NIH toolbox) from baseline
HIV-related stigma | 6, 9, 12, 24 months
  Change in HIV-related stigma (assessed using an Abbreviated Berger HIV Stigma Scale: score range 21-84, higher score indicating greater levels of stigma) from baseline
Social Connectedness | 6, 9, 12, 24 months
  Change in social connectedness (assessed using the Social Connectedness Scale: score range 20-120, higher score indicating greater sense of social connectedness and belongingness) from baseline
Sexual Behavior | 6, 9, 12, 24 months
  Change in sexual behavior of risk (assessed using questions from the Youth Risk Behavior Surveillance System) from baseline
ART Adherence | 6, 9, 12, 24 months
  Change in percentage of days, during the last 30, during which at least one dose was missed (assessed using a 30 day-recall) from baseline. Minimum= -100, maximum=100; scores above 0 indicate an improvement relative to baseline, with higher scores indicating greater improvements. Assessed among those on treatment for at least a month at enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Molly Franke, ScD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (4):
- Peru (4):
  - Hospital Nacional Arzobispo Loayza, Lima, Lima Province
  - Instituto Nacional de Salud del Nino, Breña, Lima region
  - Hospital Nacional Daniel Alcides Carrión, Callao, Lima
  - Hospital Nacional Hipólito Unanue, Lima

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code